CLINICAL TRIAL: NCT05650346
Title: Efficacy of Deep Cervical Training Combined With Mobilization Techniques on Forward Head
Brief Title: Efficacy of Deep Cervical Training Combined With Mobilization Techniques on Forward Head Posture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Egyptian Chinese University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Hamed Hasnin, Assistant Lecturer, Egyptian Chinese University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003524
Record Dates: First submitted 2022-11-23; First posted 2022-12-14 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Forward Head Posture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group ( Deep Cervical Training ) (Active Comparator)
  Interventions: Other: Deep Cervical Training
- Experimental group I (Deep cervical training + Upper cervical mobilization group) (Experimental)
  Interventions: Other: Deep Cervical Training; Other: Deep cervical training + Upper cervical mobilization group
- Experimental group II (Deep cervical training + Upper thoracic mobilization group) (Experimental)
  Interventions: Other: Deep Cervical Training; Other: Deep cervical training + Upper thoracic mobilization group

INTERVENTIONS:
Other: Deep Cervical Training — The Cranio cervical flexion exercise will be performed with the patient in supine crook lying with the neck in a neutral position (no pillow) such that the line of the face is horizontal and a line bisecting the neck longitudinally is horizontal to the testing surface. The uninflated pressure sensor will be placed behind the neck so that it abutted the occiput and is inflated to a stable baseline pressure of 20 mm Hg, a standard pressure sufficient to fill the space between the testing surface and the neck but not push the neck into a lordosis. the patient attempted to sequentially target five, 2-mm Hg progressive pressure increases from the baseline of 20 mm Hg to a maximum of 30 mm Hg as well as to maintain a isometric contraction at the progressive pressures as an endurance task.
Other: Deep cervical training + Upper cervical mobilization group — 1. the patient in supine crook lying with the neck in a neutral position.The uninflated pressure sensor will be placed behind the neck so that it abutted the occiput and is inflated to a stable baseline pressure of 20 mm Hg, a standard pressure sufficient to fill the space between the testing surface and the neck but not push the neck into a lordosis. the patient attempted to sequentially target five, 2-mm Hg progressive pressure increases from the baseline of 20 mm Hg to a maximum of 30 mm Hg
  2. The therapist will cover the rear of the cervical part of the participant with his right hand for stabilization, and will place his thumb and index fingers on the atlas of the participant. To conduct the atlanto-occipital mobilization, the therapist will place his left hand at the right side of the participant and at the same time will place his fifth finger under the occipital area and will pull the participant's head toward his trunk.
  Arms: Experimental group I (Deep cervical training + Upper cervical mobilization group)
Other: Deep cervical training + Upper thoracic mobilization group — 1. The Cranio cervical flexion exercise will be performed with the patient in supine crook lying with the neck in a neutral position (no pillow) such that the line of the face is horizontal and a line bisecting the neck longitudinally is horizontal to the testing surface. The uninflated pressure sensor will be placed behind the neck so that it abutted the occiput and is inflated to a stable baseline pressure of 20 mm Hg, a standard pressure sufficient to fill the space between the testing surface and the neck but not push the neck into a lordosis. the patient attempted to sequentially target five, 2-mm Hg progressive pressure increases from the baseline of 20 mm Hg to a maximum of 30 mm Hg as well as to maintain a isometric contraction at the progressive pressures as an endurance task.
  2. The participants will be placed in the prone position and the therapist will stand facing the joint where the mobilization will be applied to improve the extension of the upper thoracic spine (T1-2).
  Arms: Experimental group II (Deep cervical training + Upper thoracic mobilization group)

SUMMARY:
To investigate the efficacy of adding cervical & thoracic spinal mobilization techniques to deep cervical training compared to deep cervical training alone on Pain, Neck functional ability, Craniovertebral angle.

ELIGIBILITY:
Inclusion Criteria:

* The craniovertebral angle is less than 50 degrees.
* Age ranges from 18 to 25 years old.
* Forward head is associated with neck pain.

Exclusion Criteria:

A history of any of the following conditions:

* Previous surgery regarding the spine or shoulders.
* Vertebral fractures regarding the cervical spine or the skull.
* Positive neurological signs or evidence of spinal compression
* headaches prior to the onset of neck pain and without cervical origin
* Inner ear or vestibular Problems
* Whiplash Injuries

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-01-10 (Estimated); Primary Completion 2023-02-20 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral Angle | One Month
  The CVA was formed at the intersection of the horizontal line, which passed through the back and the line, which joined the tragus of the ear and the back. The Patient Will Be In Standing Position and the image will be taken from the lateral view then the image will be inserted to IMAGEJ Software To Measure The Angle
Deep Neck Core Strength | One Month
  The the patient in supine crook lying with the neck in a neutral position. The uninflated pressure sensor will be placed behind the neck so that it abutted the occiput and is inflated to a stable baseline pressure of 20 mm Hg.The movement will perform gently and slowly as a head nodding action (as if saying "yes"). The Cranio cervical flexion exercise the activation and endurance of the deep cervical flexors in progressive inner range positions as the patient attempted to sequentially target five, 2-mm Hg progressive pressure increases from the baseline of 20 mm Hg to a maximum of 30 mm Hg as well as to maintain a isometric contraction at the progressive pressures as an endurance task.

CONTACTS AND LOCATIONS:
Locations (1):
- The Egyptian Chinese University, Cairo, Egypt